CLINICAL TRIAL: NCT03894852
Title: SRSF2 Gene Mutation in Patients With Therapy Related Myelodysplastic Syndromes / Acute Myeloid Leukemia
Brief Title: SRSF2 Gene Mutation in Patients With t-MDS/AML
Status: Completed | Type: Observational
Sponsor: Zeinab Albadry Mohammed Zahran (Other)
Responsible Party: Sponsor-Investigator, Zeinab Albadry Mohammed Zahran, Assistant lecturer,Clinical Pathology Departement,Faculty of Medicine, Assiut University, Assiut University
Organization: Assiut University (Other)
Other Study IDs: SRSF2 mutation in t-MDS/AML
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Therapy Related Myelodysplastic Syndrome and Therapy Related Acute Myeloid Leukemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AML: cases with denovo AML and t-AML
  Interventions: Diagnostic Test: PCR and cytogenetics
- MDS: cases with denovo MDS and t-MDS
  Interventions: Diagnostic Test: PCR and cytogenetics

INTERVENTIONS:
Diagnostic Test: PCR and cytogenetics — detection of SRSF2 gene mutation and cytogenetic studies

SUMMARY:
* To detect SRSF2 gene mutation by polymerase chain reaction (PCR) in the two types of t-MDS/AML which recognized in the WHO classification.
* Association between SRSF2 gene mutation and the presence of other cytogenetic abnormalities in the two types of t-MDS/AML which recognized in the WHO classification, e.g. (Loss of chromosome 7 or del(7q), del(5q), isochromosome 17q, recurrent balanced chromosomal translocations involving chromosomal segments 11q23 (KMT2A, previously called MLL) or 21q22.1 (RUNX1), and PML-RARA).
* Relationship between SRSF2 gene mutation and cumulative dose, dose intensity, time of exposure and prognostic criteria (disease free survival, overall survival and disease course).

DETAILED DESCRIPTION:
Therapy-related myeloid neoplasms (t-MNs) are a group of hematologic diseases that arise after chemotherapy and/or radiation therapy for a previous cancer or rarely autoimmune diseases.

The revised 2016 World Heath Organization (WHO) classification defines t-MN as a subgroup of acute myeloid leukemia (AML) comprising myelodysplastic syndrome (t-MDS), acute myeloid leukemia (t-AML), and myelodysplastic/myeloproliferative neoplasms (t-MDS/MPN) .

Two forms of t-MN have been recognized. Alkylating agent/radiation-related t-MN usually appears 4 to 7 years, which is frequently associated with unbalanced chromosomal abnormalities involving chromosomes 5 and/or 7, as well mutations or loss of TP53 ( tumor protein 53).

In contrast, a combination of different topoisomerase II inhibitor-related t-MNs is associated with a high incidence of recurrent balanced translocations involving chromosomal segments 11q23 (KMT2A), 21q22 (RUNX1), and PML-RARA [1].

T-MNs are characterized by a subset of molecular mutations including SRSF2, SF3B1, U2AF1, ZRSR2, ASXL1, STAG2, and TP53.

RNA splicing is a process that produces mature mRNAs by excising introns and splicing exons from pre-messenger RNA. The spliceosome mutations induce an abnormally spliced mRNA species and compromising hematopoiesis.

One of the potential candidate genes involved in the RNA splicing pathway is serine and arginine rich splicing factor 2 (SRSF2). SRSF2, located on chromosome 17q25.1, and plays a role in preventing exon skipping, confirming the accuracy of splicing and regulating alternative pre-mRNA splicing. Many studies have already reported the potential prognostic value of SRSF2 mutations, which have an adverse prognostic impact on survival and disease progression.

Somatic mutations recently identified in patients with de novo AML and MDS, such as those of epigenetic regulators, spliceosome machinery and SETBP1, are rare, with the exception of SRSF2.

TP53 mutations have been associated to the occurrence of cytogenetic abnormalities and poor response to chemotherapy that are typical of t-MN.

On the other hand, several studies have shown that the presence of isochromosome 17q i(17q) abnormality is associated with wild-type TP53 and mutations in SETBP1 and SRSF2.

Also, somatic loss of one copy of the long arm of chromosome 7 del(7q) is associated with unfavorable prognosis and can co-occur with the SRSF2 mutation in patients with MDS and AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myelodysplastic syndromes (MDS), who fulfill the WHO criteria.
* Patients with acute myeloid leukemia (AML), who fulfill the WHO criteria.
* Patients must start therapy (cytotoxic agents and/or ionizing radiotherapy) before beginning of the study, with a documented history of a benign or malignant condition for which they had received therapy prior to the diagnosis of MDS or AML.

Exclusion Criteria:

* Patients not fulfill the WHO criteria for diagnosis of MDS and AML.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cases diagnosed therapy related MDS/AML admitted to department of Clinical Pathology, in the south Egypt cancer institute and Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2019-06-02 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
SRSF2 gene mutation detection in t-MDS/AML. | about 2 years
  Detect SRSF2 gene mutation by polymerase chain reaction (PCR) in the two types of t-MDS/AML which recognized in the WHO classification.

SECONDARY OUTCOMES:
Cytogenetic analysis (FISH) of patient with t-MDS/AML. | about 2 years
  Cytogenetic analysis (FISH), e.g. (Loss of chromosome 7 or del(7q), del(5q), lsochromosome 17q, recurrent balanced chromosomal translocations involving chromosomal segments 11q23 (KMT2A, previously called MLL) or 21q22.1 (RUNX1), and PML-RARA) in the two types of t-MDS/AML which recognized in the WHO classification.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Abdel-Aal Jad Elrab, Professor, Study Director — Clinical pathology Department, Faculty of Medicine, Assiut University; Sahar Abdullah El-Gammal, Assistant Professor, Principal Investigator — Clinical pathology Department, Faculty of Medicine, Assiut University; Madleen Adel Attia, Assistant Professor, Principal Investigator — Clinical pathology Department, Faculty of Medicine, Assiut University
Locations (2):
- Egypt (2):
  - Assiut, Asyut
  - Zeinab Albadry Mohammed Zahran, Asyut

REFERENCES:
- [Background] Fianchi L, Criscuolo M, Fabiani E, Falconi G, Maraglino AME, Voso MT, Pagano L. Therapy-related myeloid neoplasms: clinical perspectives. Onco Targets Ther. 2018 Sep 17;11:5909-5915. doi: 10.2147/OTT.S101333. eCollection 2018. PMID 30271175
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Sella T, Stone RM. The impact of new drugs for breast and ovarian cancer on the occurrence of therapy-related myeloid neoplasms: Understanding the baseline incidence. Gynecol Oncol. 2018 Nov;151(2):187-189. doi: 10.1016/j.ygyno.2018.10.013. No abstract available. PMID 30384959
- [Background] Hoskins AA, Moore MJ. The spliceosome: a flexible, reversible macromolecular machine. Trends Biochem Sci. 2012 May;37(5):179-88. doi: 10.1016/j.tibs.2012.02.009. Epub 2012 Apr 3. PMID 22480731
- [Background] Boultwood J, Dolatshad H, Varanasi SS, Yip BH, Pellagatti A. The role of splicing factor mutations in the pathogenesis of the myelodysplastic syndromes. Adv Biol Regul. 2014 Jan;54:153-61. doi: 10.1016/j.jbior.2013.09.005. Epub 2013 Sep 15. PMID 24080589
- [Background] Maciejewski JP, Padgett RA. Defects in spliceosomal machinery: a new pathway of leukaemogenesis. Br J Haematol. 2012 Jul;158(2):165-173. doi: 10.1111/j.1365-2141.2012.09158.x. Epub 2012 May 18. PMID 22594801
- [Background] Armstrong RN, Steeples V, Singh S, Sanchi A, Boultwood J, Pellagatti A. Splicing factor mutations in the myelodysplastic syndromes: target genes and therapeutic approaches. Adv Biol Regul. 2018 Jan;67:13-29. doi: 10.1016/j.jbior.2017.09.008. Epub 2017 Sep 22. PMID 28986033
- [Background] Fabiani E, Falconi G, Fianchi L, Criscuolo M, Ottone T, Cicconi L, Hohaus S, Sica S, Postorino M, Neri A, Lionetti M, Leone G, Lo-Coco F, Voso MT. Clonal evolution in therapy-related neoplasms. Oncotarget. 2017 Feb 14;8(7):12031-12040. doi: 10.18632/oncotarget.14509. PMID 28076841
- [Background] Visconte V, Tabarroki A, Zhang L, Hasrouni E, Gerace C, Frum R, Ai J, Advani AS, Duong HK, Kalaycio M, Saunthararajah Y, Sekeres MA, His ED, Shetty S, Rogers HJ, Tiu RV. Clinicopathologic and molecular characterization of myeloid neoplasms harboring isochromosome 17(q10). Am J Hematol. 2014 Aug;89(8):862. doi: 10.1002/ajh.23755. Epub 2014 May 16. No abstract available. PMID 24796269
- [Background] Meggendorfer M, Bacher U, Alpermann T, Haferlach C, Kern W, Gambacorti-Passerini C, Haferlach T, Schnittger S. SETBP1 mutations occur in 9% of MDS/MPN and in 4% of MPN cases and are strongly associated with atypical CML, monosomy 7, isochromosome i(17)(q10), ASXL1 and CBL mutations. Leukemia. 2013 Sep;27(9):1852-60. doi: 10.1038/leu.2013.133. Epub 2013 Apr 30. PMID 23628959
- [Background] Papapetrou EP. Patient-derived induced pluripotent stem cells in cancer research and precision oncology. Nat Med. 2016 Dec 6;22(12):1392-1401. doi: 10.1038/nm.4238. PMID 27923030
- [Background] Kanagal-Shamanna R, Bueso-Ramos CE, Barkoh B, Lu G, Wang S, Garcia-Manero G, Vadhan-Raj S, Hoehn D, Medeiros LJ, Yin CC. Myeloid neoplasms with isolated isochromosome 17q represent a clinicopathologic entity associated with myelodysplastic/myeloproliferative features, a high risk of leukemic transformation, and wild-type TP53. Cancer. 2012 Jun 1;118(11):2879-88. doi: 10.1002/cncr.26537. Epub 2011 Oct 28. PMID 22038701